CLINICAL TRIAL: NCT05686733
Title: Pre-SEAL™IT: Saccular Endovascular Aneurysm Lattice System First In Human Interventional Trial
Acronym: Pre-SEAL™IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galaxy Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0068
Record Dates: First submitted 2022-12-30; First posted 2023-01-17 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Aneurysms Saccular; Aneurysm, Ruptured; Aneurysm
MeSH Terms: conditions — Aneurysm; Aneurysm, Ruptured

STUDY DESIGN:
Intervention Model Description: First In Human (FIH), prospective, single-arm, multicenter, interventional study. Patients presenting with evidence of a single unruptured or ruptured aneurysm requiring treatment will be enrolled into the study and treated using the SEAL™ System.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (The SEAL™ Saccular Endovascular Aneurysm Lattice System) (Other): First In Human (FIH), prospective, single-arm, multicenter, interventional study.
  Interventions: Device: SEAL Device

INTERVENTIONS:
Device: SEAL Device — Endovascular treatment of target aneurysm using the Saccular Endovascular Aneurysm Lattice (SEAL) device.

SUMMARY:
To establish the preliminary safety and effectiveness of the SEAL™ Endovascular Aneurysm Lattice System for the treatment of saccular intracranial aneurysms.

The data from this study will be used to support:

1. EU CE Mark labelling
2. US FDA Investigational Device Exemption (IDE) approval support of PMA approval.

DETAILED DESCRIPTION:
First In Human (FIH), prospective, single-arm, multicenter, interventional study. Patients presenting with evidence of a single unruptured or ruptured aneurysm requiring treatment will be enrolled into the study and treated using the SEAL™ System.

Immediate post-procedure angiographic findings, clinical presentation, safety, and imaging follow-up for each subject will be collected at 24 hours, 3 (MRA), 6, 12 and 24-months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 80 years of age at the time of screening
2. Evidence of a single unruptured aneurysm requiring treatment. If there is evidence of an additional aneurysm requiring treatment, the secondary aneurysm must also be treatable using a SEAL™ System Device, either during a single procedure or consecutive procedures.

   In these instances, no additional implanted devices are permissible except for as medically required for patient safety.
   1. Ruptured aneurysms may be included according the following criteria: The subject is neurologically stable with a Hunt and Hess scale of 3 or less at the time of treatment
   2. Modified Disability Scale (mRS) of ≤2 prior to presentation or rupture
3. The index intracranial aneurysm (IA) to be treated must include the following features:

   1. Aneurysm features suitable for endovascular treatment with an intrasaccular device per the treating interventionist.
   2. Saccular morphology
   3. Located at a bifurcation, terminus, or sidewall in the anterior or posterior circulation
   4. 3mm-25mm in dome diameter
   5. Narrow or wide-neck aneurysm with neck size ≥ 4mm or Dome-to-Neck (DN) ratio < 2
4. Aneurysm treatment does not require the preplanned use of any additional implanted devices
5. Subject is able to maintain compliance with all aspects of screening, evaluation, treatment, and post-procedure follow-up schedule
6. Baseline mRS of 0-1 for unruptured cases
7. Ability to obtain written informed consent from subject prior to the initiation of any study procedures
8. Subject has been approved for inclusion by Galaxy Therapeutics INC. clinical affairs team.

Exclusion Criteria:

1. Aneurysm features unsuitable for endovascular treatment with an intrasaccular device such as fusiform, dissecting pseudo aneurysm, or mycotic aneurysm.
2. Aneurysms smaller than 3mm and larger than 25mm in dome diameter.
3. Inability to access target aneurysm with microcatheter due to intracranial atherosclerosis, vessel tortuosity or poor aneurysm angle take-off.
4. Presence of vascular disease or other vascular abnormality that could prohibit access to index aneurysm such carotid stenosis or diminished caliber of the target artery.
5. Proximal vessel tortuosity or morphology that could prohibit access to target aneurysm
6. Clinical, angiographic, or CT evidence of CNS arterial vasculitis, moyamoya disease, intracranial tumor (except small meningioma), or any other intracranial vascular malformations
7. Patients with high risk for recurrent ischemic stroke due to previous history of intracranial ischemic stroke symptoms such as transient ischemic attacks (TIAs), minor, or major strokes within the past 60 days
8. Patients with hemodynamic or medical compromise due to medical comorbidities such as severe unstable congestive heart failure (ejection fraction <30%) or severe COPD requiring home oxygen.
9. Modified Rankin Scale (mRS) score of ≤ 2 prior to presentation or acute rupture (as applicable)
10. SAH from non-index aneurysm or any other intracranial hemorrhage within the past 60 days
11. Target aneurysm has been previously treated and contains devices, implants, or coils that could interfere with correct SEAL™ device placement.
12. Subject is pregnant or a lactating female (For females of child-bearing potential, a positive pregnancy test within 7 days of the day of procedure or refusal to use a medically accepted method of birth control for the duration of the study.
13. Currently on anticoagulation therapy or has a known blood dyscrasia, coagulopathy, or hemoglobinopathy
14. Hypersensitivity that cannot be medically controlled to any component of the SEAL™ System, procedural materials, or medications commonly used during the procedure
15. Currently enrolled in another investigational study or post-market study that could affect the safety and efficacy of aneurysm treatment or interfere with the study follow- up schedule
16. Presence of an acute life-threatening illness requiring treatment
17. Life-expectancy of < 5 years
18. Subject has an uncontrolled co-morbid medical condition, including mental health issues, that would adversely affect participation in the study
19. Subject is a prisoner or member of other vulnerable population

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Procedure through 12 Months
  Subject Safety will be considered a failure upon meeting any of the following primary safety criteria:
  * Any stroke within 72 hours of the procedure or discharge home (if earlier) that results in an increase of 4 or more points on the National Institute of Health Stroke Scale
  * Major ipsilateral stroke within 72 hours post-procedure or discharge home (if earlier) to 12-months following treatment
  * New subarachnoid hemorrhage related to target aneurysm within 72 hours post-procedure or discharge home (if earlier) to 12-months following treatment
  * Death due to neurologic cause related to aneurysm treated from Procedure to 12-months following treatment
Primary Efficacy Endpoint | Procedure through 12 Months
  Proportion of subjects with aneurysm occlusion adjudicated by independent core lab based on satisfaction of the following 3 criterion:
  * WEB-IT Occlusion Scale I and II (WOS) post-implantation, at 6 months, and at 12 months
  * Raymond Roy Scale I (RRS) post-implantation, at 6 months, and at 12 months
  * Technical success defined as the proportion of subjects in whom a SEAL™ System was successfully delivered and deployed at the target aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Boris Pabón, MD, Principal Investigator — Angiosur
Locations (1):
- Clinicas Las Americas, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No